CLINICAL TRIAL: NCT03673969
Title: Mini Gastric Bypass vs Roux enY Gastric Bypass
Acronym: MGB vs RYGB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to progress the study
Sponsor: Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0945 2018 NCTS
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Gastric Bypass
Keywords: Mini Gastric Bypass; Roux En-Y Gastric Bypass; Bariatric surgery; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will not know the arm prior to surgery, but will be made aware of it afterward
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGB (Active Comparator): Mini gastric bypass
  Interventions: Procedure: Gastric bypass
- Roux enY gastric bypass (Active Comparator): Roux enY gastric bypass
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: Gastric bypass — Surgical method of gastric bypass

SUMMARY:
The primary aim of this research project is to assess the safety and efficacy of the MGB operation in the UK

DETAILED DESCRIPTION:
The main aim of this project is to develop an ideal bariatric/metabolic surgery operation.

The ideal features are highly safe operation, revisable, reversible, extremely effective, short operative time, short hospital stay, cost-effective, no long-term complications and acceptable to the patients.

Mini Gastric Bypass/One Anastomosis Gastric Bypass MGB/OAGB is relatively a new bariatric /metabolic surgery operation that is increasing in popularity and currently more than 60,000 operations are performed worldwide. Only 125 MGB operations are published from UK.

No previous RCT to date in the UK to test the new operation although RCT was done in Taiwan 2005 and showed that MGB is not inferior to the Roux EnY Gastric Bypass RYGB. This research project is assessing the outcomes of this operation and opening the doors to understand its effects and how it works compared to the standard RYGB. The possible development in the project is to study the hormonal changes after the MGB.

ELIGIBILITY:
Inclusion Criteria:

* They have a BMI of 40 kg/m2 or more, or between 35 kg/m2 and 40 kg/m2 and other significant disease (for example, type 2 diabetes or high blood pressure) that could be improved if they lost weight.
* All appropriate non-surgical measures have been tried but the person has not achieved or maintained adequate, clinically beneficial weight loss.
* The person has been receiving or will receive intensive management in a tier 3 service.
* The person is generally fit for anaesthesia and surgery.
* The person commits to the need for long-term follow-up

Exclusion Criteria:

* Not meeting the eligibility criteria
* Under 18s

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Excess weight loss | 2 years post surgery
  Amount of weight lost

SECONDARY OUTCOMES:
Type 2 diabetes remission | 6 months, 2 years, 5 years and 10 years
  Type 2 diabetes remission
Morbidity | 6 months, 2 years, 5 years and 10 years
  Morbidity
Mortality | 6 months, 2 years, 5 years and 10 years
  Mortality
Operative time | 6 months, 2 years, 5 years and 10 years
  Operative time
Length of stay | 6 months, 2 years, 5 years and 10 years
  Length of stay
Readmission rate | 6 months, 2 years, 5 years and 10 years
  Readmission rate
Lipid profile | 6 months, 2 years, 5 years and 10 years
  Lipid profile
Malnutrition | 6 months, 2 years, 5 years and 10 years
  Malnutrition
Liver failure | 6 months, 2 years, 5 years and 10 years
  Liver failure
Gastro-oesophageal reflux | 6 months, 2 years, 5 years and 10 years
  Gastro-oesophageal reflux
Upper GI cancer | 6 months, 2 years, 5 years and 10 years
  Upper GI cancer
Diarrhoea | 6 months, 2 years, 5 years and 10 years
  Diarrhoea

CONTACTS AND LOCATIONS:
Locations (1):
- Doncaster & Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Final report and findings will be appropriately disseminated following completion of the study